CLINICAL TRIAL: NCT06907433
Title: Evaluation of the Effects of Rigid Taping and Kinesiotaping on Pain, Joint Mobility and Disability in Patients with Sacroiliac Joint Dysfunction: a Randomized Controlled Trial
Brief Title: Kinesiotaping and Rigid Taping in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, MD., Ufuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09-02
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kinesiotaping group (Active Comparator)
  Interventions: Other: Rigid taping; Other: Exercise
- rigid taping group (Active Comparator)
  Interventions: Other: Kinesiotaping; Other: Exercise
- exercise group (Active Comparator)
  Interventions: Other: Kinesiotaping; Other: Rigid taping

INTERVENTIONS:
Other: Kinesiotaping — The lymphatic correction technique described by Kase for use in sacroiliac sprains or inflammations was used in KT of the dysfunctional sacroiliac joint. While the patient is standing with the spine in a neutral position, the base part of the fan-shaped cut Kinesio tape will be attached approximately 2-3 inches (approximately 5-8 cm) above the dysfunctional sacroiliac joint. Then, the patient is asked to lean forward and rotate in the opposite direction to the dysfunctional side. The tail parts of the fan-shaped tape are passed downward and inward at a 45-degree angle over the sacroiliac joint and attached to the superior edge of the gluteus maximus. The base of another kinesio tape was attached approximately 2-3 inches (approximately 5-8 cm) below the dysfunctional sacroiliac joint, the tails of the fan-shaped tape were passed upward and inward at a 45-degree angle over the sacroiliac joint and attached approximately to the upper edge of the PSIS.
  Arms: exercise group; rigid taping group
Other: Rigid taping — The technique specified in the study by Allah et al. was taken as a reference for RT of the dysfunctional sacroiliac joint. Patients were placed in a lateral position on their healthy side, with the affected side uppermost, hip flexed to 45 degrees, and the femur in a neutral position. The rigid tape was attached to the anterior superior iliac spine of the upper hip and pulled tight, and attached linearly to the posterior superior iliac spine. Another piece was attached between the same points, but in a curved shape with the opening facing downward.
  Arms: Kinesiotaping group; exercise group
Other: Exercise — Patients in all 3 groups were shown an exercise program by a physiotherapist that included lumbopelvic stabilization, flexibility and strengthening exercises for the low back and hip, and were asked to apply the exercise program for 15 days by providing visual material showing the exercises.
  Arms: Kinesiotaping group; rigid taping group

SUMMARY:
Objective: To evaluate the effects of rigid-taping and kinesiotaping (lymphatic correction) on pain, joint mobility and disability in patients with sacroiliac joint dysfunction (SIJD).

Methods: A total of 84 patients with unilateral SJID were included in this randomized controlled study. Patients were divided into kinesiotaping (KT) (n=28), rigid-taping (RT) (n=28) and control (n=28) groups. Pain levels at rest and during movement with visual analog scale (VAS) (0-10 cm), Oswestry Disability Index (ODI), mobility and pain provocation tests were recorded on days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-50 years
* patients who had subacute and chronic (lasting longer than 1 month), mechanical type low back and/or hip pain thought to be due to unilateral SIJD (spreading between 3 cm above and 10 cm below the posterior superior iliac spine, not extending above the 5th lumbar vertebra)
* patients who had at least 3 positive results out of 6 pain provocation tests for the sacroiliac joint.

Exclusion Criteria:

* the presence of known infectious, inflammatory, tumoral and advanced degenerative diseases that may cause low back pain, pain referred from abdominal or pelvic organs, history of spine or hip fracture/surgery,
* presence of nerve root involvement findings,
* presence of pregnancy, presence of inflammatory pathology in routine blood tests seen at the examination application
* presence of inflammatory or advanced degenerative changes in the sacroiliac joint in imaging methods,
* presence of findings suggesting bilateral sacroiliac joint dysfunction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
pain intensity with movement and at rest on a 0-10 cm visual analog scale (VAS) scale (0=no pain, 10=unbearable pain) | 15 days
Oswestry Disability Index | 15 days

SECONDARY OUTCOMES:
The number of positive mobility test | 15 days
The number of positive pain provacation test | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided